CLINICAL TRIAL: NCT00396903
Title: Evaluation of a Standard Epidural Catheter During Clinical Practice
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: O-H-0403
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Patients Scheduled for Epidural Anaesthesia
Keywords: Anaesthetic techniques; epidural catheters; paraesthesia; side effects.
MeSH Terms: conditions — Paresthesia | interventions — Catheters

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: catheter

SUMMARY:
During the insertion of epidural catheters several complications can occur, including transient paraesthesia and inadvertent venous cannulation.

Reported incidences for paraesthesia vary widely between about 0.2% and 50% in different articles, depending on the catheter (catheter material, soft-tipped or firm-tipped catheter), the applied technique (lumbar or thoracic epidural anesthesia, depth of catheter insertion), the approach (midline or paramedian) and the included patients (obstetrical or non-obstetrical). Furthermore, the inconsistent definition of "paraesthesia" makes it difficult to compare the results of different studies. Paraesthesia are not supposed to lead to permanent neurological sequelea, but are unpleasant and perturbing sensations for the patient.

For inadvertent venous cannulation during epidural catheter placement, incidences between 1% and 14% have been reported. As for the paraesthesia rate, catheter material, technique, approach and included patients are determinants for the incidence of vessel puncture.

Main objective of this study is to determine the incidence of paraesthesia with this catheter.

Secondary objectives are to record

* the frequency of inadvertent venous cannulation
* difficulties involved in insertion and removal of the catheter
* data on additional complications
* data for the evaluation of handling characteristics

DETAILED DESCRIPTION:
Study design

This study is a prospective, uncontrolled, open, non-randomised study ("Observational Study") with a CE-certified medical device.

Patients

Information and consent Information of the procedure and oral consent of epidural anaesthesia for the surgery is obtained as usual. Oral consent for data collection has to be obtained. No randomisation or blinding is performed and no non-standard procedures are necessary.

Inclusion criteria 100 patients scheduled for Epidural Anaesthesia will be included in this study. Eligible patients are ASA class I-III, between 18 and 75 years of age and are scheduled for EA, with or without general anaesthesia.

Exclusion criteria Anamnestic exclusion criteria are all contraindications for epidural anaesthesia (e.g. neurological deficit, skin infection of the puncture site, diseases leading to neurological impairment such as diabetes, coagulation impairment). Non-competent and non-cooperative patients as well as pregnant and breast-feeding women are also to be excluded. Same applies for patients with medicament- and drug abuse or problems in communication or those participating in parallel in another clinical study with experimental drugs or devices.

Randomisation and Blinding No randomization is required. An independent observer who is not performing the epidural will record occurrence, incidence and intensity of paraesthesia.

Definition of the main and the secondary criteria

Main criteria

- Frequency of paraesthesia during catheter insertion

Secondary criteria

* Frequency of inadvertent venous cannulation (aspiration of blood)
* Intensity of paraesthesia (VAS)

  * description: - pain
* electric shock
* burning sensation
* shooting effect
* motor reactions (right/left)
* discomfort
* others
* Frequency and kind of difficulties during insertion of the catheter (rating of "easiness of insertion": 0 = no resistance, 1 = minor difficulties, 2 = serious difficulties, 3 = impossible)
* Facultative: Documentation of paraesthesia/difficulties during catheter removal at 48 hours after surgery (or earlier, if appropriate)

Concomitant parameters

* Patient data (age, height, weight, sex, diagnosis, kind of intervention, ASA class, relevant co-diagnosis, relevant co-medication)
* Epidural anaesthesia and -analgesia related data

  • Data that relate to the description of the puncture process and method chosen in case of difficulties during puncture, catheter insertion and removal
  * Level of sensory blockade
  * Indwelling time of epidural catheter by recording the time of insertion
  * Dose/kind of anaesthetic used for epidural anaesthesia, type of general anaesthesia if relevant
  * Kind of analgesia done by epidural catheter
  * Adequacy of epidural anaesthesia (yes / no)
  * Further complications/side effects related to epidural anaesthesia/analgesia (i.e. dural puncture, haematoma, etc)
* Judgement of the anaesthesiologist concerning handling features (0 = no resistance, 1 = minor difficulties, 2 = serious difficulties)
* Catheter damages

ELIGIBILITY:
Inclusion Criteria:

* scheduled for Epidural Anaesthesia
* ASA class I-III
* between 18 and 75

Exclusion Criteria:

* contraindications for epidural anaesthesia
* Non-competent and non-cooperative
* pregnant and breast-feeding women
* medicament- and drug abuse or problems in communication
* participating in parallel in another clinical study with experimental drugs or devices

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-04; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Frequency of paraesthesia during catheter insertion

CONTACTS AND LOCATIONS:
Overall Officials: Marco Marcus, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands

REFERENCES:
- [Result] Bouman EA, Gramke HF, Wetzel N, Vanderbroeck TH, Bruinsma R, Theunissen M, Kerkkamp HE, Marcus MA. Evaluation of two different epidural catheters in clinical practice. narrowing down the incidence of paresthesia! Acta Anaesthesiol Belg. 2007;58(2):101-5. PMID 17710897